CLINICAL TRIAL: NCT04180007
Title: Evaluating the Safety and Efficacy of Radioactive Iodine (RAI) Treatment of Metastatic and Advanced Differentiated Thyroid Cancers by Pretreatment With Apatinib for the Neoadjuvant Regimen
Brief Title: Study of Neoadjuvant Regimen for Radioactive Iodine Treatment of Metastatic and Advanced Differentiated Thyroid Cancers
Acronym: APT-01
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, FengWang, Director of Nuclear Medicine, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: wangfeng-Apatinib-001
Record Dates: First submitted 2019-11-24; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Thyroid; Metastasis; Apatinib
MeSH Terms: conditions — Thyroid Diseases; Neoplasm Metastasis | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant arm (Experimental): Patients receive Apatinib orally qd up to 12 wk.
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — 500 mg Apatinib given orally once a day for 12 wk prior to RAI (131I) treatment.

SUMMARY:
The purpose of this study is to determine Safety and Efficacy of Radioactive Iodine (RAI) Treatment of Metastatic and Advanced Differentiated Thyroid Cancers by Pretreatment With Apatinib for the Neoadjuvant Regimen

DETAILED DESCRIPTION:
This study is design to prospectively investigate the safety and efficacy of apatinib in downsizing primary tumors and metastatic lesions in patients with metastatic and advanced differentiated thyroid cancers before RAI Treatment.

Standard treatment of thyroid cancer includes thyroidectomy, RAI treatment, and levothyroxine replacement therapy. Before RAI treatment, L-thyroxin replacement therapy should be stopped to induce TSH elevation, thereby promoting the intake of radioactive iodine in residual or metastatic lesions. However, the process of withdrawing L-thyroxin for 4-6 weeks might promote the progression of the tumor. The main hypothesis is that the use of tyrosine kinase inhibitor will reduce the tumor proliferation or metastasis rate of patients before RAI Treatment.

Apatinib is a tyrosine kinase inhibitor that selectively inhibits the vascular endothelial growth factor receptor-2. This is a single-institution, single-arm phase 2 clinical trial. Patients will receive axitinib 500mg qd for up to 12 week. Patients then will receive RAI Treatment. If the severe adverse effects discontinued study treatment prior to 12 week, the patient may also receive subsequent RAI treatment at the time of suspension. The follow-up period was followed up to assess safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

1. The patient volunteers and signs an informed consent form.
2. age ≥18 and <99 years old;
3. Diagnosed as differentiated thyroid cancer (DTC) by histopathology;
4. surgically inoperable and/or recurrent/metastatic differentiated thyroid cancers;
5. Did not receive molecular targeting treatment; Prior RAI therapy is allowed if > 3 months prior to initiation of therapy on this protocol and evidence of progression (as defined above) has been documented in the interim.
6. There must be at least one measurable lesion (according to RECIST v1.1);
7. Physical condition ECOG PS: 0-2;
8. Expected survival time ≥ 3 months;
9. Laboratory tests meet the following criteria: Bone marrow function: absolute count of blood neutrophils (ANC) ≥1.5×109/L; platelet (PLT)≥100×109/L; hemoglobin (HB)≥90g/L; Liver function: alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ULN*2.5
10. Well controlled blood pressure prior to study entry.
11. At least one or more hypermetabolic lesions other than the neck on 18F-FDG PET scans

Exclusion Criteria:

1. Anaplastic thyroid carcinoma, thyroid lymphoma, mesenchymal tumors of the thyroid, metastases to the thyroid;
2. Previous treatment with chemotherapy for anti-thyroid cancer (allowing low-dose chemotherapy for radiation sensitization) or treatment with thalidomide or its derivatives;
3. Previous treatment with VEGFR-TKI small molecule drugs within 1 month, such as vandetanib, cabozantinib, lenvatinib, sunitinib, sorafenib, etc.;
4. Major surgery within 4 weeks prior to enrollment, or received anti-thyroid cancer radiotherapy;
5. Severe cardiovascular disease, including hypertension (BP≥140/90mmHg) uncontrolled by medical treatment, unstable angina, history of myocardial infarction, congestive heart failure>NYHA II, Marked baseline prolongation of QT/corrected QT (QTc) interval;
6. Severe infection requires intravenous antibiotic, antifungal or antiviral treatment;
7. Active hemoptysis (bright red blood of at least one-half teaspoon) in the 28 days prior to study entry;
8. Suffering from mental illness, poor compliance;
9. Pregnant women will be ineligible; breast feeding should be discontinued if the mother is treated with Apatinib;
10. Embolization and bleeding occurred within 4 weeks before enrollment;
11. Patient with a risk of gastrointestinal bleeding; abnormal coagulation function (INR > 1.5, APTT > 1.5 × ULN);
12. Arteriovenous thrombosis such as cerebrovascular accidents, deep vein thrombosis, and pulmonary embolism within 12 months prior to screening;
13. A variety of factors that affect the absorption of oral medications (such as inability to swallow, nausea and vomiting, chronic diarrhea and intestinal obstruction)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-04-10 (Actual); Primary Completion 2020-04-10 (Estimated); Study Completion 2020-05-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 4 month
  Number of patients achieving a complete response (CR) or partial response (PR) by Response Evaluation Criteria (RECIST v1.1 criteria) in Solid Tumors.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Time interval from start to 3 months after completion of the therapy
  This study will utilize the CTCAE (NCI Common Terminology Criteria for Adverse Events) Version 4.0 for toxicity and Serious Adverse Event reporting
Change From Baseline in Serum Thyroglobulin Levels After Treatment With RAI (131I) | Baseline, 4 weeks, 12 weeks and 1 month after RAI

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, PhD MD, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jingsu, China

REFERENCES:
- [Derived] Shi L, You Q, Wang J, Wang H, Li S, Tian R, Yao X, Wu W, Zhang L, Wang F, Lin Y, Li S. Antitumour effects of apatinib in progressive, metastatic differentiated thyroid cancer (DTC). Endocrine. 2022 Oct;78(1):68-76. doi: 10.1007/s12020-022-03113-9. Epub 2022 Jun 29. PMID 35767182